CLINICAL TRIAL: NCT02768805
Title: Immunogenicity, Safety, and Tolerability of a Plant-Derived Quadrivalent VLP Influenza Vaccine in Adults 18-64 Years of Age
Brief Title: Immunogenicity of a Quadrivalent Virus-Like Particles (VLP) Influenza Vaccine in Healthy Adults
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medicago (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CP-Q14VLP-009
Record Dates: First submitted 2016-04-01; First posted 2016-05-11 (Estimated); Last update posted 2020-06-11 (Actual); Status verified 2020-06

CONDITIONS: Virus Diseases; RNA Virus Infections; Respiratory Tract Diseases; Respiratory Tract Infections
Keywords: Influenza; Human; RNA Virus Infections; Immunologic; Immunogenic Factors; Physiological Effects of Drug; Virus Diseases; Orthomyxoviridae Infections; Infection
MeSH Terms: conditions — Virus Diseases; RNA Virus Infections; Respiratory Tract Diseases; Respiratory Tract Infections; Influenza, Human; Orthomyxoviridae Infections; Infections

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 15 µg/strain of Quadrivalent VLP Vaccine (Experimental)
  Interventions: Biological: 15 µg/strain of Quadrivalent VLP Vaccine
- 30 µg/strain of Quadrivalent VLP Vaccine (Experimental)
  Interventions: Biological: 30 µg/strain of Quadrivalent VLP Vaccine
- 15 µg/strain of the licensed quadrivalent vaccine (Active Comparator)
  Interventions: Biological: 15 µg/strain of the licensed quadrivalent vaccine

INTERVENTIONS:
Biological: 15 µg/strain of Quadrivalent VLP Vaccine — Single dose of non-adjuvanted Quadrivalent VLP Vaccine
  Arms: 15 µg/strain of Quadrivalent VLP Vaccine
Biological: 30 µg/strain of Quadrivalent VLP Vaccine — Single dose of non-adjuvanted Quadrivalent VLP Vaccine
  Arms: 30 µg/strain of Quadrivalent VLP Vaccine
Biological: 15 µg/strain of the licensed quadrivalent vaccine — Single dose of the licensed quadrivalent vaccine
  Other Names: FluLaval® Tetra; FluLaval® Quadrivalent
  Arms: 15 µg/strain of the licensed quadrivalent vaccine

SUMMARY:
This Phase 2 Quadrivalent VLP Vaccine study is intended to replicate and extend the immunogenicity and safety results obtained in earlier Phase 1-2 and Phase 2 studies. The study is being conducted to demonstrate that the immunogenicity profile of the Quadrivalent VLP Vaccine meets the US Center for Biologics Evaluation and Research (CBER) licensure criteria. The study will also help to define the optimal dose, establish potential competitive advantages, and support the design of future studies.

DETAILED DESCRIPTION:
This randomized, observer-blind, multicenter, Phase 2 study will be conducted at multiple sites across the United States and Canada.

The influenza strain composition of the Quadrivalent VLP Vaccine used in this study includes 2 influenza A virus strains (A/California/7/2009 [H1N1] and A/Switzerland/9715293/2013 [H3N2]) and 2 influenza B virus strains (B/Phuket/3073/2013 [Yamagata lineage] and B/Brisbane/60/2008 [Victoria lineage]), based on the 2015-2016 recommended World Health Organization (WHO) strains for vaccination in the Northern hemisphere.

Approximately 900 healthy subjects will be randomized in a 1:1:1 ratio to 1 of 3 parallel treatment groups. Subjects in each group will be stratified into 2 age strata: 18 to 49 years and 50 to 64 years in a 2:1 ratio.

Subjects will receive one intramuscular (IM) injection of their assigned vaccine:

* 15 µg/strain of Quadrivalent VLP Vaccine, or
* 30 µg/strain of Quadrivalent VLP Vaccine, or
* 15 µg/strain of the licensed and commercially available quadrivalent vaccine FluLaval® Tetra.

Subjects will participate in this study for approximately 8 months, during which 5 visits will be scheduled, and phone contact will be made on Day 1, Day 8, and every 2 months thereafter for up to 6 months post-Day 21 visit (Day 201). Safety laboratory assessments will be performed at Screening, on Day 3 and within 48 hours of Day 3 results availability, for grade 3 or grade 4 abnormalities or if deemed necessary by the investigator or early termination.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must be able to read, understand, and sign the informed consent form (ICF); complete study-related procedures; and communicate with the study staff at visits and by phone.
2. Subjects are considered by the Investigator to be reliable and likely to cooperate with the assessment procedures and be available for the duration of the study.
3. Male and female subjects must be 18 to 64 years of age, inclusive, at Screening (Visit 1).
4. Subjects have a body mass index (BMI) of ≥ 18.0 and ≤ 32.4 kg/m2 at Day 0.
5. Subjects must be in good general health prior to study participation (no more than 30 days prior to study vaccine administration) with no clinically relevant abnormalities that could jeopardize subject safety or interfere with study assessments as assessed by the Principal Investigator or sub-Investigator (thereafter referred as Investigator) and determined by medical history, physical examination, biochemistry, hematology, and urinalysis. Note: Subjects with a pre-existing chronic disease will be allowed to participate if the disease is stable and, according to the Investigator's judgment, the condition is unlikely to confound the results of the study or pose additional risk to the subject by participating in the study. Stable disease is generally defined as no new onset or exacerbation of pre-existing chronic disease 6 months prior to immunization. Based on the Investigator's judgment, a subject with more recent stabilization of a disease could also be eligible.
6. Female subjects must have a negative serum pregnancy test result at Screening (Visit 1) and a negative urine pregnancy test at Randomization prior to immunization.
7. Female subjects of childbearing potential must use an effective method of contraception for 1 month prior to immunization and agrees to continue employing adequate birth control measures for at least 60 days post-immunization. Moreover, she must have no plan to become pregnant for at least 2 months post-immunization. Abstinent subjects should be asked what method(s) they would use, should their circumstances change, and subjects without a well-defined plan should be excluded.

   The following relationship or methods of contraception are considered to be effective:
   * Hormonal contraceptives (e.g., injectable, topical [patch], or estrogenic vaginal ring);
   * Intra-uterine device with or without hormonal release;
   * Male partner using a condom plus spermicide or sterilized partner (at least 1 year prior to immunization);
   * Credible self-reported history of heterosexual abstinence until at least 60 days postimmunization;
   * Female partner.
8. Non-childbearing females are defined as:

   * Surgically-sterile (defined as bilateral tubal ligation, hysterectomy or bilateral oophorectomy performed more than 1 month prior to immunization); or
   * Post-menopausal (absence of menses for 24 consecutive months and age consistent with natural cessation of ovulation).

Exclusion Criteria:

Subjects who meet any of the following criteria will be excluded from participating in this study:

1. According to the Investigator's opinion, history of significant acute or chronic, uncontrolled medical or neuropsychiatric illness. "Uncontrolled" is defined as:

   * Requiring a new medical or surgical treatment within one month prior to study vaccine administration;
   * Requiring a change in medication dosage during one month prior to study vaccine administration due to uncontrolled symptoms or drug toxicity, or for chronic diseases, significant change in medication dosage within 6 months prior to study vaccine administration based upon the investigator's judgment (elective dosage adjustments in stable subjects are acceptable).
2. Any medical or neuropsychiatric condition or any history of excessive alcohol use or drug abuse which, in the Investigator's opinion, would render the subject unable to provide informed consent or unable to provide valid safety observations and reporting.
3. Any autoimmune disease other than hypothyroidism on stable replacement therapy or any confirmed or suspected immunosuppressive condition or immunodeficiency including known or suspected human immunodeficiency virus (HIV), Hepatitis B or C infection, or the presence of lymphoproliferative disease.
4. Administration or planned administration of any non-influenza vaccine within 30 days prior to randomization up to blood sampling at Day 21. Immunization on an emergency basis will be evaluated case-by-case by the Investigator.
5. Administration of any adjuvanted or investigational influenza vaccine within 1 year prior to randomization or planned administration prior to the completion of Day 201.
6. Administration of any 'standard', non-adjuvanted influenza vaccine (e.g., live attenuated trivalent/quadrivalent inactivated influenza vaccine Intranasal or split trivalent/quadrivalent inactivated influenza vaccine by either intradermal or intramuscular [IM] route) within 6 months prior to randomization and up to completion of Day 21 visit.
7. Use of any investigational or non-registered product within 30 days or 5 half-lives, whichever is longer, prior to randomization or planned use during the study period. Subjects may not participate in any other investigational or marketed drug study while participating in this study until Day 201 visit.
8. Treatment with systemic glucocorticoids at a dose exceeding 10 mg of prednisone per day, or equivalent for more than 7 consecutive days or for 10 or more days in total, within one month of study vaccine administration, any other cytotoxic or immunosuppressant drug, or any immunoglobulin preparation within 3 months of vaccination and until the completion of Day 21 visit. Low doses of nasal or inhaled glucocorticoids are allowed. Topical steroids are permitted.
9. Any significant disorder of coagulation including treatment with warfarin derivatives or heparin. Persons receiving prophylactic anti-platelet medications (e.g., low-dose aspirin [no more than 325 mg/day]), and without a clinically apparent bleeding tendency are eligible. Subjects treated with new generation drugs that do not increase the risk of intramuscular bleeding (e.g., clopidogrel) are also eligible.
10. History of allergy to any of the constituents of the Quadrivalent VLP vaccine (including H1N1, H3N2, B/Bris, and B/Phuket), to any components of the licensed quadrivalent vaccine, or tobacco allergy.
11. History of anaphylactic allergic reactions to any food, medication, or bee sting.
12. Any history of serious asthma (e.g., status asthmaticus, hospitalization for asthma control) or recurrent asthma episodes requiring medical attention in the last 3 years (≥ 1 episode/year)
13. Continuous use of antihistamines in the last 4 weeks prior to immunization or use of antihistamines 48 hours prior to study immunization.
14. Use of prophylactic medications (e.g. acetaminophen/paracetamol, aspirin, naproxen, or ibuprofen) within 24 hours of randomization to prevent or pre-empt symptoms due to vaccination. Subject discovered to have taken a prophylactic medication within the 24 hours prior to planned randomization must be delayed until at least the 24 hours period is met.
15. Have a rash, dermatological condition, tattoos, muscle mass, or any other abnormalities at injection site that may interfere with injection site reaction rating.
16. Have received a blood transfusion within 90 days prior to study vaccination.
17. If female subject, have a positive or doubtful pregnancy test result prior to immunization or lactating females.
18. Have abnormal vital signs defined as: systolic Blood Pressure (BP) > 140 mmHg and/or diastolic BP ≥ 90mmHg, heart rate ≤ 45 beats/min and ≥ 100 beats/min. Even if one or more vital signs are out of the acceptable ranges, a subject may still be included in the study based on Investigator's judgment (e.g. a resting heart rate ≤ 45 in highly-trained athletes). Presence of any febrile illness (including oral temperature (OT) ≥ 38.0 ˚C within 24 hours prior to immunization). Such subjects may be re-evaluated for enrolment after resolution of illness.
19. Cancer or treatment for cancer within 3 years of study vaccine administration. Persons with a history of cancer who are disease-free without treatment for 3 years or more are eligible. Persons with treated and uncomplicated basal cell carcinoma of the skin are eligible. Person with non-treated, non-disseminated local prostate cancer are eligible.
20. Identified as an Investigator or employee of the Investigator or clinical site with direct involvement in the proposed study, or identified as an immediate family member (i.e., parent, spouse, natural or adopted child) of the Investigator or employee with direct involvement in the proposed study or any employees of Medicago.
21. Subject with a history of Guillain-Barre Syndrome.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 900 (Actual)
Dates: Start 2016-03-02; Primary Completion 2016-05-17 (Actual); Study Completion 2016-11-26 (Actual)

PRIMARY OUTCOMES:
Immunogenicity assessed by the geometric mean titers (GMT) of hemagglutination inhibition (HI) antibody against the homologous influenza strains | 21 days after injection
  Immunogenicity will be assessed by the geometric mean titers (GMT) of hemagglutination inhibition (HI) antibody against the homologous influenza strains

SECONDARY OUTCOMES:
Immunogenicity assessed by GMT of HI antibody against heterologous strains | 21 days after injection
  Immunogenicity will be assessed by GMT of HI antibody against heterologous strains
Immunogenicity assessed by GMT of microneutralization (MN) antibody against homologous and heterologous strains | 21 days after injection
  Immunogenicity will be assessed by GMT of microneutralization (MN) antibody against homologous and heterologous strains
Immunogenicity assessed by GMT of single radial hemolysis (SRH) antibody against homologous and heterologous strains | 21 days after injection
  Immunogenicity will be assessed by GMT of single radial hemolysis (SRH) antibody against homologous and heterologous strains
Immunogenicity assessed by cell-mediated immune (CMI) response against homologous and heterologous strains | 21 days after injection
  Immunogenicity will be assessed by cell-mediated immune (CMI) response against homologous and heterologous strains
Incidence of Solicited Local and Systemic Reactions | 21 days after injection
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | 21 days after injection
Incidence of Abnormal Clinical Laboratory Tests | 3 days after injection

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Lachance, MD, Principal Investigator — Centre de Recherche St-Louis, Quebec, Canada; Marc Dionne, MD, Principal Investigator — Équipe de recherche en vaccination du CHU de Québec-Université Laval (CHU), Quebec, Canada; Michael Libman, MD, Principal Investigator — McGill University Health Center - Vaccine Study Center (MUHC), Montreal, Canada; Trevor Wesson, MD, Principal Investigator — Diex Research Montreal, Montreal, Canada; Ginette Girard, MD, Principal Investigator — Diex Research Sherbrooke, Sherbrooke, Canada; Deepen Patel, MD, Principal Investigator — Topstone Research, Toronto, Canada; Diane Krieger, MD, Principal Investigator — Miami Research Associates (MRA), Miami (FL), USA; David Seiden, MD, Principal Investigator — Broward Research Group (BRG), Hollywood (FL), USA; Suchet R Patel, MD, Principal Investigator — Regional Clinical Research (RCR), Endwell (NY), USA
Locations (9):
- United States (3):
  - Broward Research Group (BRG), Hollywood, Florida
  - Miami Research Associates (MRA), South Miami, Florida
  - Regional Clinical Research (RCR), Endwell, New York
- Canada (6):
  - Topstone Research, Toronto, Ontario
  - Diex Research Montreal, Montreal, Quebec
  - McGill University Health Center - Vaccine Study Center (MUHC), Pierrefonds, Quebec
  - Diex Research Sherbroooke, Sherbrooke, Quebec
  - Équipe de recherche en vaccination du CHU de Québec-Université Laval (CHU), Québec
  - Centre de Recherche St-Louis, Québec

IPD SHARING:
Plan to Share IPD: No